CLINICAL TRIAL: NCT06945276
Title: A Phase 1 Study to Evaluate Relative Bioavailability and Food Effect of an ALG-097558 Tablet Formulation and the Drug-Drug Interaction Potential of ALG-097558 and Its Metabolite ALG-097730 in Healthy Volunteers
Brief Title: Phase 1 Study on Bioavailability, Food Effect, and Drug-Drug Interaction of ALG-097558 Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0026
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04-18

CONDITIONS: COVID-19
Keywords: ALG-097558; Dabigatran; Drug-Drug Interaction; Healthy Subjects; Interventional; Itraconazole; SARS-CoV-2; Tablet Formulation
MeSH Terms: conditions — COVID-19 | interventions — Dabigatran; Itraconazole

STUDY DESIGN:
Intervention Model Description: Part A and B are single group. Part C is crossover.
Who Masked: Participant
Masking Description: Participants are only masked in Part A. Parts B and Part C are open label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part A Arm (Experimental): A single-blind oral placebo dose will be administered on Day 1. On Day 2, an open-labeled single oral dose of 300 mg of ALG-097558 will be administered as a spay-dried dispersion (SDD) tablet, followed by a washout period of at least 2 days. On Day 4-10 participants will receive a daily oral dose of Itraconazole 200 mg. A single oral dose of matching placebo (SDD tablet) for ALG-097558 will be given on Day 6, and a single oral dose of 300 mg of ALG-097558 SDD tablet will be given on Day 7. (N=12)
  Interventions: Drug: ALG-097558; Drug: Itraconazole; Other: Placebo
- Part B Arm (Experimental): A single oral dose of 75 mg of dabigatran will be administered on Day 1, in a fasted stated, followed by a washout period of at least 3 days. Participants will then receive multiple oral doses of 600 mg of ALG-097558 Q12H as a spray-dried dispersion (SDD) tablet on Days 4-5, in a fasted state. A single oral dose of 75 mg of dabigatran will be given on Day 5, in a fasted state. (N=24)
  Interventions: Drug: ALG-097558; Drug: Dabigatran
- Part C Sequence 1 Arm (Experimental): A single oral dose of 600 mg of ALG-097558, in a spray-dried dispersion (SDD) tablet will be administered in the fasted state, followed by a 3-day washout period. On Day 4, a single oral dose of 600 mg of ALG-097558, in a conventional tablet will be administered in the fasted state, followed by another 3-day washout period. On Day 7, a single oral dose of 600 mg of ALG-097558, in a conventional tablet will be administered in the fed state. (N=5)
  Interventions: Drug: ALG-097558
- Part C Sequence 2 Arm (Experimental): A single oral dose of 600 mg of ALG-097558, in a conventional tablet will be administered in the fasted state, followed by a 3-day washout period. On Day 4, a single oral dose of 600 mg of ALG-097558 in a conventional tablet will be administered in the fed state, followed by another 3-day washout period. On Day 7, a single oral dose of 600 mg of ALG-097558, in a spray-dried dispersion (SDD) tablet will be administered in the fasted state. (N=5)
  Interventions: Drug: ALG-097558
- Part C Sequence 3 Arm (Experimental): A single oral dose of 600 mg of ALG-097558, in a conventional tablet will be administered in the fed state, followed by a 3-day washout period. On Day 4, a single oral dose of 600 mg of ALG-097558 in a spray-dried dispersion (SDD) tablet will be administered in the fasted state, followed by another 3-day washout period. On Day 7, a single oral dose of 600 mg of ALG-097558, in a conventional tablet will be administered in the fasted state. (N=5)
  Interventions: Drug: ALG-097558

INTERVENTIONS:
Drug: ALG-097558 — A selective, reversible, and potent inhibitor of the SARS-CoV-2 3CLpro with pan-coronavirus activity
Drug: Dabigatran — A direct thrombin inhibitor approved for the treatment and prevention of blood clots to reduce the risk of stroke
  Arms: Part B Arm
Drug: Itraconazole — A substrate and strong dual inhibitor of CYP3A4/P-glycoprotein (P-gp)
  Arms: Part A Arm
Other: Placebo — Placebo
  Arms: Part A Arm

SUMMARY:
The aim of this multi-part Phase 1 study is to evaluate the drug-drug interaction (DDI) potential of ALG-097558 via co-administration with a P-gp substrate (dabigatran) and a CYP3A4 inhibitor/P-gp inhibitor (itraconazole). In addition, this study will evaluate the relative bioavailability and food effect of a new tablet formulation for ALG-097558.

This study consists of 3 parts, all conducted in healthy volunteers (HV). Study Parts A and B are designed to assess the perpetrator or victim DDI risk of ALG-097558 mediated by CYP/P-gp interactions in healthy adult subjects. Part A will evaluate the potential impact of itraconazole, a CYP3A potent inhibitor, while Part B will investigate the potential impact of ALG-097558 (perpetrator) on dabigatran etexilate, a P-gp transporter substrate. Study Part C is designed to study the bioavailability of a new formulation of the ALG-097558 tablet and the food effect on this tablet.

This study has one primary objective for each part of the study. For Part A: to evaluate the effect of a CYP3A4 inhibitor/Pg-p inhibitor, itraconazole, on the pharmacokinetics (PK) of ALG-097558 and the metabolite, ALG-097730. For Part B: to evaluate the effect of multiple doses of ALG-097558 on the pharmacokinetics of a P-gp substrate, dabigatran. For Part C: to evaluate the relative bioavailability of 2 different tablet formulations of ALG-097558 and effect of food on the pharmacokinetics of ALG-097558 and the metabolite, ALG-097730.

DETAILED DESCRIPTION:
The aim of this multi-part Phase 1 study is to evaluate the drug-drug interaction (DDI) potential of ALG-097558 via co-administration with a P-gp substrate (dabigatran) and a CYP3A4 inhibitor/P-gp inhibitor (itraconazole). In addition, this study will evaluate the relative bioavailability and food effect of a new tablet formulation for ALG-097558.

This study consists of 3 parts, all conducted in healthy volunteers (HV). As ALG-097558 is a substrate of CYP3A4 and P-gp transporters, any concomitant administration of an inhibitor or inducer drug may alter its exposures. Part A will evaluate the potential impact of itraconazole, a CYP3A potent inhibitor, on the ALG-097558 (victim) systemic exposure in a single group, partially-blinded study. Part B will investigate the potential impact of ALG-097558 (perpetrator) on dabigatran etexilate, a P-gp transporter substrate in a single group, open-label study. Study Part C is designed to study the bioavailability of a new formulation of the ALG-097558 tablet and the food effect on this tablet in an open-label, randomized, crossover study.

This study has one primary objective for each part of the study. For Part A: to evaluate the effect of a CYP3A4 inhibitor/Pg-p inhibitor, itraconazole, on the pharmacokinetics (PK) of ALG-097558 and the metabolite, ALG-097730. For Part B: to evaluate the effect of multiple doses of ALG-097558 on the pharmacokinetics of a P-gp substrate, dabigatran. For Part C: to evaluate the relative bioavailability of 2 different tablet formulations of ALG-097558 and effect of food on the pharmacokinetics of ALG-097558 and the metabolite, ALG-097730.The study has secondary objectives for each part of the study as well. For Part A: to evaluate the safety and tolerability of single doses of ALG-097558 in HV participants when administered as monotherapy or in combination with itraconazole. For part B: to evaluate the safety and tolerability and PK of multiple doses of ALG-097558 in HV participants when administered alone or in combination with dabigatran. For part C: to evaluate the safety and tolerability of single doses of ALG-097558 in HV participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is able to read the written informed consent, states willingness to comply with all study procedures, and is anticipated to be available for all study visits.
2. Male or female adults between 18 and 65 years of age, inclusive.
3. Female participants must either be postmenopausal*, permanently sterile**, or of childbearing potential with acceptable birth control methods***.

   *Postmenopausal: a postmenopausal state is defined as no menses for at least 12 months without an alternative medical explanation, confirmed by a high follicle-stimulating hormone (FSH) level in the postmenopausal range at screening. NOTE: If there is a question about menopausal status in women on hormone replacement therapy (HRT), the woman will be required to use one of the protocol-defined non-estrogen-containing hormonal highly effective contraceptive methods if she wishes to continue HRT during the study.

   **Permanently sterile: methods include hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal ligation, or bilateral tubal occlusion.
   * Women of childbearing potential (WOCBP): are only eligible if they and any non-sterile, male sexual partners agree to use protocol-defined highly effective (dependent or independent) contraceptive therapy, from the start of dosing until at least 90 days after the last dose. Acceptable method of contraception, hormonal contraceptives (e.g., oral, injectable, implantable, insertable, and transdermal patch), intrauterine device (with or without hormones), or double-barrier method (e.g., condom and spermicide) for 30 days prior to Screening, during the study, and for 90 days following the last administration of investigational product (IP). WOCBP must also agree to refrain from egg donations during the study and for at least 90 days following the last administration of IP.
4. Male participants who must agree to wear a condom with spermicide during sexual intercourse.*

   *These contraceptive measures must be implemented, at a minimum, from the start of dosing until at least 90 days after the last dose. Male volunteers must agree not to donate sperm during the study and for 90 days following the last administration of IP.
5. Participants must have a body mass index (BMI) of 18.0 to 32.0 kg/m^2, extremes included.
6. Participants must be nonsmokers for at least 3 months prior to randomization/enrollment.
7. Participants must have a 12-lead electrocardiogram (ECG) that considered in an acceptable range for inclusion.*

   *Criteria includes: heart rate between 40 and 100 beats per minute [bpm], extremes included; QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) </= 450 ms (males) or </= 470 ms (females); QRS interval </=120 ms; PR interval >/=110 to </=220 ms; and in addition to fulfilling the above ECG criteria, ECG morphology must have no clinically significant abnormalities observed.

   NOTE: Retesting of an apparently exclusionary ECG will be allowed once without prior approval from the Sponsor (following ECG collections described in Section 8.3.4). Participants with a retest ECG without clinically significant abnormalities as per this inclusion criterion may be included.
8. Participants must be deemed to be in good overall health by the Investigator on the basis of a medical evaluation* performed at Screening.

   *Medical evaluation that includes the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs, and the results of blood chemistry, blood coagulation and hematology tests, and urinalysis.
9. Subject must be willing and able to adhere to the Prohibited Medication requirements and Special Precautions as specified in the protocol.

Exclusion Criteria:

1. Participants with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose risk in administering study drug to the subject.* *Additionally illnesses that could prevent, limit, or confound the protocol specified assessments or study results' interpretation. This may include, but is not limited to, renal, cardiac, vascular, pulmonary, gastrointestinal, hepatologic, endocrine, neurologic, dermatologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances.
2. Participants with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome or clinical evidence at screening of significant or unstable cardiac disease.*

   *Risk factors for Torsade de Pointes syndrome include hypokalemia and family history of long QT syndrome. Clinical evidence of cardiac disease include angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, clinically significant ECG abnormalities, moderate to severe valvular disease or uncontrolled hypertension. Evidence of heart block or bundle branch block, inclusive of first-degree AV block and incomplete bundle branch block, on ECG is also exclusionary.
3. Participants with a history of clinically significant drug allergy such as, but not limited to, sulfonamides or drug allergy witnessed in previous studies with experimental drugs.
4. Participants with a recent (within 1 year of randomization/enrollment) history of use of amphetamines, barbiturates, narcotic or other drugs of abuse/recreational drug use.*

   *Use of these drugs under physician supervision (e.g., prescription narcotics for known pain disorder) are not exclusionary. Cannabis use is also not exclusionary unless detected at screening or Day -1 (Exclusion Criteria 7).
5. Excessive use of alcohol defined as regular consumption of >/=14 standard drinks/week .*

   *For current definition of a standard drink, refer to the National Institute on Alcohol Abuse and Alcoholism website.
6. Unwilling to abstain from alcohol use for 1 week prior to start of study through end of study follow up.
7. Positive results for urine drug screen for barbiturates, opiates, amphetamines, methadone, cocaine, benzodiazepines, or cannabinoids, alcohol or cotinine test at screening and Day - 1.
8. Participants with current viral infections.*

   *Viral infections include the following:
   * Hepatitis A virus infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]).
   * Hepatitis B infection defined as presence of HBsAg or HBV core antibody.
   * Hepatitis C virus (HCV) infection (confirmed by HCV antibody and/or HCV RNA). Participants who have been treated and achieved sustained virologic response >/=6 months prior to screening with HCV RNA < Lower limit of quantitation (LLOQ), target not detected, remain eligible.
   * Hepatitis E virus: Anti-HEV IgM-positive and/or detectable HEV RNA level (only applies to participants with history of living or traveling to an HEV epidemic area within 90 days of screening).
   * Human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening.
   * Acute infection at the time of randomization/enrollment. If an acute infection is considered resolved prior to randomization/enrollment, the subject remains eligible.
9. Male participants who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug.
10. Women who are breastfeeding or planning to breastfeed throughout the duration of the study.
11. Use of any medications (prescription and Over-the-counter (OTC)), vitamins, and/or herbal supplements* within 1 week (or 5 half-lives, whichever is longer) prior to the first dose of study drug.

    *Exception of contraceptives and OTC doses of ibuprofen or acetaminophen of up to 3 doses per week
12. Use of prohibited medications (as described in Section 6.8.1) within 14 days (or 5 half-lives, whichever is longer) prior to the first dose of study drug.
13. Consumption of grapefruit, grapefruit juice, and Seville oranges within 7 days prior to first study drug administration.
14. Consumption of apple or orange juice, citrus fruits, vegetables from the mustard green family*, and charbroiled meats within 7 days prior to first study drug administration.

    *Examples are kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard.
15. Consumption of any food or drink/beverage containing quinine (e.g., tonic, bitter lemon, bitter alcoholic beverages containing quinine) within 24 hours prior to study drug administration.
16. Participants having received an investigational agent within 30 days (or 5 half-lives, whichever is longer) prior to screening.
17. Participants currently participating in another clinical or medical interventional research study.
18. Participants with any >/=Grade 1 laboratory result that is considered clinically significant by the Investigator at screening. (Grade 1 laboratory result that is not clinically significant is allowed.)
19. Clinically significant abnormal vital signs* (evaluated in the supine position after at least 5 minutes of rest), confirmed with retesting after at least 5 minutes of additional rest.

    *Abnormal vital signs are based on the following criteria:
    * Systolic blood pressure: <90 or >145 mmHg
    * Diastolic blood pressure: <50 or >95 mmHg
    * Pulse rate: <45 or >100 beats per minute
    * Temperature: <36.1 degrees Celsius or >38.0 degrees Celsius
20. Physical examination findings that are considered clinically significant per study principal investigator and/or study physician and likely to adversely impact study conduct and/or interpretation are exclusionary.
21. Participants who had major surgery (e.g., requiring general anesthesia) within 12 weeks before screening, planned during the study, or within 4 weeks after the last dose of study drug.*

    *This includes participants who will not have fully recovered from surgery by the time the participant is expected to participate in the study. NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate.
22. Participants with renal dysfunction*

    *Includes estimated creatinine clearance <80 mL/min/1.73 m^2 at screening or Day -1, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. CKD-EPI should not be corrected for participants of African ancestry.
23. Participants with alanine aminotransferase (ALT) values >1.2× upper limit of normal (ULN) at screening or Day -1.
24. Participants who donated blood or plasma recently*

    *Recently defined as within 56 days prior to screening, or loss of whole blood of more than 500 mL within 30 days prior to Day-1, or receipt of a blood transfusion within 1 year of study enrollment; receipt of Plasma 7 days prior to screening.
25. Participant is an employee of the Sponsor, the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site.* *This extends to family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity [extrapolated] (AUC0-inf) | Up to Day 10
Area under the concentration-time curve from time zero to the last measurable concentration (AUClast) | Up to Day 10
Elimination half-life (t1/2) | Up to Day 10
Initial concentration (C0) | Up to Day 10
Maximum observed concentration (Cmax) | Up to Day 10
Minimum observed concentration (Cmin) | Up to Day 10
Time of observed maximum concentration (Tmax) | Up to Day 10

SECONDARY OUTCOMES:
Incidence of adverse events | Up to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

DOCUMENTS (3):
  • Informed Consent Form: Part_A_Itraconazole (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT06945276/ICF_000.pdf
  • Informed Consent Form: Part_B_Dabigatran (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT06945276/ICF_001.pdf
  • Informed Consent Form: Part_C_ALG-097558 (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT06945276/ICF_002.pdf